CLINICAL TRIAL: NCT05056935
Title: A Randomized, Double-Blind, Placebo-Controlled Proof of Concept Study to Evaluate LB1148 for Return of Gastrointestinal Function, Decrease Post-Operative Ileus in Subjects Undergoing Elective Bowel Resection
Brief Title: Study to Evaluate LB1148 for Return of Gastrointestinal Function, Decrease Post-Operative Ileus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBS-POI-201
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Ileus
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LB1148 (Experimental): active
  Interventions: Drug: LB1148
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LB1148 — A total of 700 mL of LB1148 will be administered orally as a split dose before surgery.
  Arms: LB1148
Drug: Placebo — A total of 700 mL of placebo will be administered orally as a split dose before surgery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish preliminary evidence of the efficacy, safety, and tolerability of LB1148 for the treatment of return of gastrointestinal function and decrease Post-Operative Ileus in subjects undergoing elective bowel resection.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo an elective (non-emergent) bowel resection with or without a planned stoma via laparotomy or minimally invasive technique. This includes any subject in which a resection of the small intestine, colon, or rectum is performed for any elected indication.
2. Has been informed of the nature of the study (either the subject or their legal representative), agrees to its provisions, and has provided written informed consent.

Exclusion Criteria:

1. <18 or >80 years of age.
2. Requires emergency bowel surgery.
3. Has had 1 or more abdominal surgeries, excluding the current, for inflammatory bowel disease, including, but not limited to, inflammatory bowel disease (IBD), Crohn's Disease, or ulcerative colitis.

   Note: This does not apply to previous surgery such as hernia repair unrelated to IBD.
4. American Society of Anesthesiologists (ASA) Class 4 or 5.
5. Insulin dependent diabetes mellitus.
6. Known inability to take the study drug orally (i.e. complete small bowel obstruction).
7. Has contraindications or potential risk factors to taking tranexamic acid (TXA). These include subjects with:

   1. Known sensitivity to tranexamic acid (TXA);
   2. Recent craniotomy (past 30 days);
   3. Active cerebrovascular bleed;
   4. Active thromboembolic disease (such as deep vein thrombosis, pulmonary embolism, cerebral thrombosis, ischemic stroke, or acute coronary syndrome);
   5. Acute promyelocytic leukemia taking all-trans retinoic acid for remission induction, or
   6. Continuing use of a combined hormonal contraceptive and or combined hormonal replacement therapy (including combined hormonal pill, patch, or vaginal ring).
8. Known allergic reaction to polyethylene glycol (PEG) 4000 powder, combination formulation of polyethylene glycol (PEG) and electrolyte powder, polyethylene glycol (PEG) 3350 solution and glucose formulation.
9. Has the following risk factors for thromboembolic disease:

   1. Known medical history of congenital or acquired thrombophilia such as, but not limited to patients with:

      * Sickle cell disease;
      * Nephrotic syndrome;
      * Factor V Leiden;
      * Prothrombin gene mutation;
      * Protein C or S deficiency;
      * Antithrombin III deficiency;
      * Antiphospholipid syndrome.
   2. Stage IV malignant neoplasm;
   3. Neurologic paresis, partial paralysis, or paralysis;
   4. Pacemaker;
   5. History of pulmonary embolism, deep vein thrombosis, cerebrovascular accident, or rental venous/arterial occlusion;
10. History of or current seizure disorder.
11. Patients with myeloproliferative disorders.
12. Body Mass Index (BMI) >40.
13. Any other condition that, in the opinion of the Investigator, would preclude the subject from being an appropriate candidate for the study, including severe renal or hepatic impairment.
14. Planned treatment with alvimopan (Entereg®) during study participation period.
15. Received any other investigational therapy within 4 weeks prior to Randomization
16. Chronic opioid usage, defined by the American Pain Society as daily or near-daily use of opioids for at least 90 days.
17. Female subjects of childbearing potential with a positive urine or serum pregnancy test or who are not taking (or not willing to take) acceptable birth control measures (abstinence, intrauterine devices, contraceptive implants or barrier methods) through Day 30. Additionally, those women who are lactating and insist on breast feeding within 5 days of the last dose of study drug.
18. Known history of radiation enteritis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-08-08 (Actual)

PRIMARY OUTCOMES:
Time to reach GI-2 | within 14 days after surgery
  • GI-2 is defined as the toleration of solid food and first bowel movement.
  * Ability to tolerate a solid oral diet is defined as the time from the end of surgery (the time of last skin staple or suture is placed by surgeon) to the time a patient finishes first solid meal that requires chewing and no significant nausea or vomiting for 4 hours after solid meal).
  * First bowel movement is defined as the time from the end of surgery to the first passage of stool.

SECONDARY OUTCOMES:
Time to reach GI-3 | within 14 days after surgery
  • GI-3 is defined as the toleration of solid food and either first flatus or bowel movement.
Nausea Verbal Rating Scoring Scale | within 14 days after surgery
  • To assess the nausea and ability to tolerate food
Number of days in the hospital | within 14 days after surgery
  • Length of Stay (number of days in the hospital, evaluated in hours) will be measured by time to
  * Discharge order is written,
  * Actual discharge, and
  * Standard discharge criteria

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - General Hospital of Xuzhou Mining Group, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Ningbo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No